CLINICAL TRIAL: NCT03747705
Title: A Controlled Trial for Prevention of Loss of the Effect of Epilepsy Drugs
Brief Title: Trial for Epilepsy Patients Non-responsive to AEDs Using Medical App
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Tahel Ilan Ber (Industry)
Responsible Party: Sponsor-Investigator, Tahel Ilan Ber, CMO, Oberon Sciences LTD
Organization: Oberon Sciences LTD (Industry)
Other Study IDs: Os-001
Record Dates: First submitted 2018-11-17; First posted 2018-11-20 (Actual); Last update posted 2019-02-05 (Actual); Status verified 2019-02

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: An App for reminding patients to take their medication — Open-label, single-center study, up to 20 adults (>18) male and female with, intractable epilepsy, on stable doses of antiepileptic drugs (AEDs), will participate in a 4-week observation period during which no change in the drugs is permitted. The patients will then begin 10-week treatment by taking their medications according to a semi-random schedule that is pre-set for them by the physician using the same drugs the patient is taking and only changing the dose and times of taking them each day while keeping the drugs within their therapeutic window. Between 6:00-22:00 During the study, patients will fill a seizure diary daily.

SUMMARY:
Trial for epilepsy patients non-responsive to AEDs, using medical app reminding patients to take their physician-prescribed medications

ELIGIBILITY:
Inclusion Criteria:

1. Patients in whom seizures are not controlled by their anti-seizure medication
2. Must have at least 2 seizures per month
3. History of any of the following seizure types: tonic, clonic, tonic-clonic in the form of partial seizures, partial seizures secondarily generalized or primary generalized, complex partial seizures and drop attacks (tonic/atonic)
4. At least four clinically countable seizures within 4 weeks of study entry [tonic, clonic, tonic-clonic in the form of partial seizures, partial seizures secondarily generalized or primary generalized and/or complex partial seizures and drop attacks (tonic/atonic)]
5. The subject to a stable regimen of 1-4 concomitant antiepileptic drugs (AEDs) for a minimum of 4 weeks prior to enrollment
6. History of treatment with at least two AEDs, including one trial of a combination of at least two concomitant drugs, without successful seizure control
7. Subjects with vagal nerve stimulation system must be in stable settings for a minimum of 6 months prior to enrollment
8. RNS deep brain stimulation or the ketogenic diet can be considered equivalent to a drug trial and must be on a stable ratio for a minimum of 3 months prior to enrollment
9. Completed seizure diary for four weeks (±3 days) prior to initiation of the dose titration period (visit 2). The subject will be considered a screen failure if seizure diary was not appropriately completed
10. Anti-epileptic drugs at stable doses for a minimum of 4 weeks prior to enrollment.

Exclusion Criteria:

1. Neurodegenerative or deteriorated neurological disease
2. Psychosis or past psychotic event and/or anxiety disorder
3. Current or history of drug abuse/addiction
4. Abnormal creatinine
5. Any chronic ophthalmology disease
6. The subject is currently using or has used cannabis-based or synthetic cannabinoid within three months of study entry
7. Renal, hepatic [ALT/AST >2x upper limit of normal (ULN), bilirubin >2x ULN], pancreatic dysfunctions or laboratory test abnormalities, at the investigator's discretion
8. The subject is pregnant, lactating, or planning a pregnancy during the course of the study or within 3 months of study completion
9. The subject is currently enrolled in or has not yet completed a period of at least 60 days since ending another investigational device or drug trial(s)
10. Unable to comply with study visits/requirements
11. Diagnosis of Dravet Syndrome, Lennox-Gastaut syndrome, or any other congenital or childhood syndrome will be excluded completely from this trial
12. Female subjects who are pregnant will be excluded from the study. If a female subject is able to become pregnant, she will be given a serum pregnancy test before entry into the study. Female subjects will be informed not to become pregnant while on trial. Female subjects must tell the investigator and consult an obstetrician or maternal-fetal specialist if they become pregnant during the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with drug-resistant epilepsy
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2019-03-01 (Estimated); Primary Completion 2019-11-12 (Estimated); Study Completion 2019-11-12 (Estimated)

PRIMARY OUTCOMES:
Change in seizure frequency from baseline to the seizure count evaluation period | 10 weeks

SECONDARY OUTCOMES:
Change in seizure frequency from baseline to the seizure count evaluation period | 10 weeks
Overall Quality of Life in Epilepsy-31 (QOLIE-31) Score in Patients With Baseline & at Least One Post-baseline QOLIE Assessment | 10 weeks
Changes in the Number of Anti-epileptic Drugs Prescribed | 10 weeks
Changes in Anti-Epileptic Drugs (AEDs) in patients with less than a 50% reduction in seizures | 10 weeks

REFERENCES:
- [Derived] Azmanov H, Ross EL, Ilan Y. Establishment of an Individualized Chronotherapy, Autonomic Nervous System, and Variability-Based Dynamic Platform for Overcoming the Loss of Response to Analgesics. Pain Physician. 2021 May;24(3):243-252. PMID 33988944